CLINICAL TRIAL: NCT07026344
Title: Efficacy of Rescue Stenting/Angioplasty After Failed Thrombectomy for Acute Large Intracranial Vascular Occlusion: A Multicenter, Prospective, Open-label, Endpoint-blinded, Randomized Controlled Trial
Brief Title: Efficacy of Rescue Stenting/Angioplasty After Failed Thrombectomy for Acute Large Intracranial Vascular Occlusion
Acronym: ANGEL-RESCUE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANGEL-RESCUE
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Thrombectomy; Large Intracranial Vascular Occlusion; Rescue Stenting; Randomized Controlled Trial
MeSH Terms: conditions — Ischemic Stroke | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stenting or Angioplasty Group (Experimental): If recanalization is not achieved after 3-5 attempts of thrombectomy, direct stent placement or balloon angioplasty is performed.
  Interventions: Procedure: Stent placement; Procedure: balloon angioplasty
- Continued Thrombectomy Group (Active Comparator): If recanalization is not achieved after 3-5 attempts of thrombectomy, at least one additional thrombectomy attempt is performed
  Interventions: Procedure: Continued Thrombectomy

INTERVENTIONS:
Procedure: Stent placement — For patients who fail thrombectomy, perform stent placement.
  Arms: Stenting or Angioplasty Group
Procedure: Continued Thrombectomy — For patients with failed thrombectomy, perform at least one additional thrombectomy attempt
  Arms: Continued Thrombectomy Group
Procedure: balloon angioplasty — For patients who fail thrombectomy, perform balloon angioplasty.
  Arms: Stenting or Angioplasty Group

SUMMARY:
The primary objective of this study is to evaluate whether rescue stenting therapy can improve neurological functional outcomes after failed endovascular treatment for acute ischemic stroke caused by large vessel occlusion. The study population is divided into two groups:

Stent Placement Group: If recanalization is not achieved after 3-5 attempts of thrombectomy, direct stent placement or balloon angioplasty is performed.

Continued Thrombectomy Group: If recanalization is not achieved after 3-5 attempts of thrombectomy, at least one additional thrombectomy attempt is performed.

The primary efficacy endpoint is the proportion of patients achieving a modified Rankin Scale (mRS) score of 0-2 at 90±7 days.

The safety endpoint is the incidence of symptomatic intracranial hemorrhage within 48 hours after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Pre-stroke mRS 0-1
3. Symptoms of AIS present within 24 hours of last known well time
4. Baseline NIHSS score ≥6
5. Anterior circulation: ASPECTS ≥6; Posterior circulation: pc-ASPECTS ≥6
6. Occlusion of intracranial ICA, M1 segment of MCA, V4 segment of vertebral artery, or basilar artery
7. Clinical care team intends to perform endovascular therapy (EVT)
8. Failure to achieve recanalization (eTICI 0-1) after 3 thrombectomy attempts, including: At least one contact aspiration attempt; At least one stent retriever attempt or combined approach
9. Subject or legally authorized representative can provide informed consent

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by imaging prior to randomization; or intraprocedural flat-panel CT evidence of major hemorrhage
2. Gastrointestinal or genitourinary bleeding within 30 days post-stroke onset; or major surgery within 14 days
3. Bleeding diathesis, including:Laboratory evidence of coagulopathy (PLT <100×10⁹/L, aPTT >50 sec, or INR >2.0); Direct oral anticoagulant (DOAC) use within 48 hours prior; History of heparin-induced thrombocytopenia (HIT)
4. Pregnancy or lactation at admission
5. Contraindications to:Radiographic contrast agents; Nickel, titanium, or their alloys (device-related)
6. Life expectancy <6 months
7. Pre-existing neurological/psychiatric conditions that may confound neurological assessment
8. Severe renal insufficiency:GFR <30 mL/min or Serum creatinine >220 μmol/L (2.5 mg/dL)
9. Arterial tortuosity or other vascular anomalies preventing device delivery to target vessel
10. Unlikely to complete 90-day follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with mRS 0-2 | 90±7 days
  Proportion of patients with Modified Rankin Scale (mRS) 0-2, Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.

SECONDARY OUTCOMES:
Change in NIHSS score from baseline | 36±12 hours post-randomization
  Change in National Institute of Health stroke scale score from baseline.The NIH Stroke Scale (NIHSS) score ranges from 0 to 42 points, with lower scores indicating better neurological function
Vascular recanalization rate assessed by CT/MR angiography | at 36±12 hours post-randomization
  Vascular recanalization rate assessed by CT/MR angiography
Change in infarct volume | at 7±3 days post-randomization or discharge (whichever comes first)
  Change in infarct volume
Distribution of mRS scores | 7±3 days/discharge and 90±7 days post-randomization
  Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.
Proportion of patients achieving mRS 0-1 | 90±7 days
  Proportion of patients achieving mRS 0-1
Incidence of rescue therapy | 90±7 days
  Incidence of rescue therapy
EQ-5D-5L utility score | 90±7 days
  The EuroQol 5-Dimension 5-Level Utility Score (EQ-5D-5L utility score) ranges from -0.594 to 1.000 (Chinese value set), assessing health-related quality of life, with higher scores indicating better health status.
Probability of symptomatic intracranial hemorrhage | 48 hours
  Probability of symptomatic intracranial hemorrhage
All-cause mortality | 90±7 days post-randomization
  All-cause mortality
Probability of any intracranial hemorrhage (per Heidelberg criteria) | 48 hours post-randomization
  Probability of any intracranial hemorrhage (per Heidelberg criteria)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No